CLINICAL TRIAL: NCT01946139
Title: Screening HIV-Infected Women for Anal Cancer Precursors
Brief Title: Anal HPV Tests in Screening for Cell Changes in the Anus in Patients With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AMC-084; NCI-2013-01637 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-084 (Other: AIDS - Associated Malignancies Clinical Trials Consortium); AMC-084 (Other: CTEP); R01CA163103 (NIH); U01CA121947 (NIH)
Record Dates: First submitted 2013-09-17; First posted 2013-09-19 (Estimated); Results first posted 2022-09-30 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-04

CONDITIONS: Anal Cancer; HIV Infection; Human Papilloma Virus Infection
MeSH Terms: conditions — Anus Neoplasms; HIV Infections; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Screening (HSIL detection) (Experimental): Patients undergo screening for the detection of HSIL using anal cytology, HPV hybrid capture 2, HPV mRNA assays, and OncoHealth HPVE6/E7 oncoprotein at baseline, at 6, 12, 18, and 24 months.
  Interventions: Procedure: comparison of screening methods; Other: laboratory biomarker analysis; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: comparison of screening methods — Undergo HPV screening using HC2, APTIMA and OncoHealth HPV E6/E7 assays
Other: laboratory biomarker analysis — Correlative studies
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This clinical trial studies anal human papillomavirus (HPV) tests in screening for cell changes in the anus in patients with human immunodeficiency virus (HIV). Screening tests may help doctors find cancer cells early and plan better treatment for anal cancer. Completing multiple screening tests may help find the best method for detecting cell changes in the anus.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the sensitivity and specificity of HPV testing using different methods of detection, including HPV Hybrid Capture 2 (HC2), HPV messenger ribonucleic acid (mRNA) assays (APTIMA) and OncoHealth HPV E6/E7 oncoprotein assay and whether they improve the screening performance of routine anal cytology for the detection of anal high-grade squamous intraepithelial lesions (HSIL) when measured against the gold standard, biopsy-proven HSIL.

II. To determine the prevalence and risk factors for prevalent HSIL in HIV-infected women.

III. To determine incidence and risk factors associated with anal HSIL and HPV over 2 years among HIV infected women undergoing semi-annual anal evaluations.

EXPLORATORY OBJECTIVES:

I. To evaluate the acceptability of anal cancer screening among HIV-infected women.

II. To collect data on quality of life and health care costs (including non-direct health care costs and time costs) for an economic evaluation of the cost-effectiveness of anal cancer screening strategies in HIV-positive women.

OUTLINE:

Patients undergo screening for the detection of HSIL using anal cytology, HPV hybrid capture 2, HPV mRNA assays, and OncoHealth HPVE6/E7 oncoprotein at baseline, at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive; HIV-1 infection, as documented by any federally approved, licensed HIV rapid test performed in conjunction with screening (or enzyme-linked immunosorbent assay [ELISA], test kit, and confirmed by Western blot or other approved test); alternatively, this documentation may include a record that another physician has documented that the participant has HIV infection based on prior ELISA and Western blot, or other approved diagnostic tests
* Karnofsky performance status > 70%
* Absolute neutrophil count >= 750 cells/mm^3 within 120 days of study entry
* Platelet count >= 75,000 cells/mm^3 within 120 days of study entry

Exclusion Criteria:

* Current or history of anal or perianal carcinoma
* History of anal HSIL cytology or histology
* Known permanent or irreversible bleeding disorder, or any illness that, in the opinion of the clinical investigator, would contraindicate any biopsy of the anal canal
* For women able to conceive, evidence of pregnancy by a positive urinary pregnancy test; pregnant women are excluded from enrollment in this study
* Serious medical or psychiatric illness that in the opinion of the site Investigator will interfere with the ability of the subject to give informed consent or adhere to the protocol
* Ongoing use of anticoagulant therapy other than aspirin, clopidogrel or non-steroidal anti-inflammatory drugs (NSAIDS)
* Inability to provide informed consent
* Treatment of anal and/or perianal HPV associated disease (i.e., condyloma or low-grade anal intraepithelial neoplasia [AIN]) within 4 months of study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2013-12-04 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Chiao, Principal Investigator — AIDS Associated Malignancies Clinical Trials Consortium
Locations (12):
- United States (11):
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - Ucsf Ancre, San Francisco, California
  - John H. Stroger Hospital of Cook County, Chicago, Illinois
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Weill-Cornell Medical College, New York, New York
  - Laser Surgery Care Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
- University of Puerto Rico Comprehensive Cancer Center, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- Screening (HSIL Detection): Patients undergo screening for the detection of high grade squamous intraepithelial lesions (HSIL) using anal cytology, human papillomavirus (HPV) hybrid capture 2, HPV mRNA assays, and OncoHealth HPVE6/E7 oncoprotein at baseline, at 6, 12, 18, and 24 months.
  comparison of screening methods: Undergo HPV screening using HC2, APTIMA and OncoHealth HPV E6/E7 assays
  laboratory biomarker analysis: Correlative studies
  questionnaire administration: Ancillary studies
  quality-of-life assessment: Ancillary studies
Period: Overall Study
Arm/Group | Screening (HSIL Detection)
Started | 276
Completed | 256
Not Completed | 20
Not completed — Withdrawal by Subject | 8
Not completed — ineligible | 8
Not completed — Specimens not available | 4

BASELINE CHARACTERISTICS:
Population: Participants who were entered into the AMC084 study
Arm/Group | Screening (HSIL Detection)
Number analyzed (Participants) | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 251
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 256
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51
  Not Hispanic or Latino | 199
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 168
  White | 61
  More than one race | 6
  Unknown or Not Reported | 17
Region of Enrollment [Number; unit: participants]
  United States | 256
Anal HSIL at baseline [Count of Participants; unit: Participants] | 69

OUTCOME MEASURES:

1. Primary Outcome: Specificity of Each Other Methods of HSIL Detection for APTIMA Assay
Description: Among patients who are HRA negative for HSIL, the number of participants who tested negative for HSIL on the APTIMA assay
Time Frame: at baseline
Population: Participants who were negative for HSIL on the high resolution anoscopy at baseline and who had APTIMA assay results
Measure: Count of Participants; unit: Participants
Arm/Group | Screening (HSIL Detection)
Number analyzed (Participants) | 175
Participants | 116

2. Primary Outcome: Prevalence of HSIL
Description: The prevalence of HSIL will be estimated as the proportion of women who are HRA positive for HSIL at entry and its 95% confidence interval. Logistic regression analysis will be used to evaluate the association of potential risk factors with diagnosis of HSIL.
Time Frame: at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Screening (HSIL Detection)
Number analyzed (Participants) | 256
Participants | 69

3. Primary Outcome: Sensitivity of Each of the Methods of APTIMA Assay at Baseline
Description: Among patients whose high resolution anoscopy (HRA) results were positive for HSIL and had APTIMA assays at baseline, the number whose APTIMA assay results were positive.
Time Frame: at baseline
Population: Patients whose HRA results were positive and had APTIMA results at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Screening (HSIL Detection)
Number analyzed (Participants) | 68
Participants | 50

4. Primary Outcome: Incidence of HSIL Among Women Who Were HRA Negative for HSIL at Study Entry
Description: The Poisson rate and its 95% confidence interval will be estimated from the number of HSIL cases detected divided by the cumulative years of follow-up across these cases.
Time Frame: Up to 2 years
Population: Participants who did not have HSIL at baseline based on the high resolution anoscopy (HRA) results and who had follow-up HRA results
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Screening (HSIL Detection)
Number analyzed (Participants) | 143
events per 100 person-years | 9.08 [6.09 to 13.55]

5. Secondary Outcome: Acceptability of Anal Cancer Screening
Description: Anal cancer screening is typically done using a high resolution anoscopy, a device which allows visualization of the anus. To determine if participants found anal screening acceptable, they were asked if they were at east with having a high resolution anoscopy. The results indicated the number of participants who felt at ease with having a high resolution anoscopy
Time Frame: at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Screening (HSIL Detection)
Number analyzed (Participants) | 256
Participants | 137

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Screening (HSIL Detection)
All-Cause Mortality (participants affected / at risk) | 1/256
Serious Adverse Events (participants affected / at risk) | 4/256
Other Adverse Events (participants affected / at risk) | 17/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Screening (HSIL Detection) (N=256)
Chest pain - Cardiac (Cardiac disorders) | 1
Bone infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Skin and subcutaneous tissue disorder, other (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Screening (HSIL Detection) (N=256)
Blurred vision (Eye disorders) | 1
Eye disorders, other (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 8
Anal pain (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Injury, poisoning and procedural complications, other (Injury, poisoning and procedural complications) | 1
Pregnancy, puerperium and perinatal conditions, other (Pregnancy, puerperium and perinatal conditions) | 2
Vaginal discharge (Reproductive system and breast disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures, other (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT01946139/Prot_SAP_000.pdf
  • Informed Consent Form (2014-09-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT01946139/ICF_001.pdf